CLINICAL TRIAL: NCT01226706
Title: Efficacy of Botulinum Toxin A Intradetrusor Injections for the Treatment of Non-neurogenic Urinary Urge Incontinence- A Randomized Double-Blind Control Trial
Brief Title: Efficacy of Botulinum Toxin Type A for the Treatment of Non-neurogenic Urinary Urge Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Corrine Jabs, Department Head Obstetrics & Gynecology, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB-08-04; 120486 (Registry Identifier: Health Canada)
Record Dates: First submitted 2010-10-18; First posted 2010-10-22 (Estimated); Results first posted 2017-07-03 (Actual); Last update posted 2017-07-03 (Actual); Status verified 2017-04

CONDITIONS: Urinary Urge Incontinence
Keywords: Urinary incontinence, urge; detrusor hyperreflexia; detrusor instability; non-neurogenic; Female Urogenital Diseases and Pregnancy Complications; Female Urogenital Diseases; Urologic Diseases; Urination Disorders; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive; Female Urogenital Diseases and Pregnancy Complications; Female Urogenital Diseases; Urologic Diseases; Urination Disorders; Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebos (Placebo Comparator): Placebo injected into the detrusor at Day 1,
  Interventions: Drug: Placebos
- Botulinum Toxins, Type A (Experimental): Botulinum Toxins, Type A 100U injected into the detrusor at Day 1
  Interventions: Drug: Botulinum Toxins, Type A

INTERVENTIONS:
Drug: Botulinum Toxins, Type A — Botulinum Toxins, Type A 100U injected into the detrusor at Day 1
  Arms: Botulinum Toxins, Type A
Drug: Placebos — Placebos injected into the detrusor at Day 1, followed by injection of botulinum toxin Type A 100U after 24 weeks has elapsed from previous treatment, if requested/qualified.
  Arms: Placebos

SUMMARY:
Non-neurogenic urinary urge incontinence (UUI) is a common quality of life disorder that causes people to feel an "urgent" need to urinate. Standard treatment for UUI includes behavior modification, pelvic floor exercises, anticholinergic medication, and less commonly, sacral neuromodulation. Unfortunately anticholinergic therapy is only moderately effective.

Botulinum toxin A (BTA or Botox©) may be a useful treatment in patients that do not respond to standard therapy. Botulinum toxin A has been used in other studies to improve symptoms in neurogenic urinary incontinence, and a variety of lower urinary tract disorders. BTA has been used in other studies to improve the symptoms in urinary incontinence, migraines, spinal cord injuries and a variety of lower urinary tract disorders. However, the treatment of non-neurogenic urinary urge incontinence has not been examined in a well-controlled study.

The primary purpose of this study is to determine the efficacy of botulinum toxin A (BTA) in the treatment of non-neurogenic urinary urge incontinence (UUI). The secondary objectives are to examine the side effects associated with BTA treatment and the impact this treatment has on patients' quality of life.

DETAILED DESCRIPTION:
Introduction:

Non-neurogenic urinary urge incontinence (UUI) is a common quality of life disorder that becomes more prevalent with age. It is described as a condition that causes people to feel an "urgent" need to urinate due to muscle spasms in the bladder. Factors such as infection, inflammation, strokes, and dementia can stimulate the bladder to create spasms and cause urine loss. Overactive bladder refers to the symptom complex of urinary frequency, urgency and or nocturia with or without incontinence. Overactive bladder is a disorder of the storage phase of the bladder affecting approximately 16.9% of the US women, increasing to 31% after age 75. Standard treatment for UUI includes behavior modification, pelvic floor exercises, anticholinergic medication, and less commonly, sacral neuromodulation. Unfortunately anticholinergic therapy is only moderately effective and causes bothersome side effects, particularly at higher doses. Sacral neuromodulation therapy is currently unavailable in Saskatchewan with the closest treatment centre being located in Calgary.

Botulinum toxin A (BTA or Botox©) may be a useful treatment in patients that do not respond to standard therapy. Botulinum toxin A has been used in other studies to improve symptoms in neurogenic urinary incontinence, migraines following spinal cord injuries, and a variety of lower urinary tract disorders. This product has been approved by FDA for treatments of the following conditions: two eye muscle disorders (blepharospasm and strabismus in December 1989), severe underarm sweating (primary axillary hyperhydrosis), brow furrow and frown lines (April 2002) and other cosmetic purposes (July 2004). For the treatment of UUI, BTA is injected into the detrusor muscle of the bladder which is the muscle of the bladder that squeezes urine towards the outlet. BTA has been used in other studies to improve the symptoms in urinary incontinence and a variety of lower urinary tract disorders, however, the treatment for non-neurogenic urinary urge incontinence has not been examined in a well-controlled study.

Research Purpose and Objectives:

The primary purpose of this study is to determine the efficacy of BTA in the treatment of non-neurogenic UUI. The secondary objectives are to examine the side effects associated with BTA treatment and the impact this treatment has on patients' quality of life.

Research Methods:

This study employs a 12 month, double-blinded, randomized, partial cross-over design. The first 6 months of the study, subjects will be randomized to receive either detrusor injection of BTA or a placebo injection. In the remaining six months, subjects in the control group will be offered the detrusor injection of BTA. All 36 subjects will be followed for the remaining 6 months.

Study Procedures and Protocol

Pre-injection Assessment:

The pre-injection and assessment stage includes an evaluation of the medical history and physical exam. Previous therapy and medication will be disclosed to the physician. The investigator will ensure the subject meets the inclusion criteria, has had urinalysis and a pregnancy test if under 50 years old.

Day of the Procedure:

On the day of the surgery, the study pharmacist will randomize subjects using a random numbers table. The study doctor, nurses, and subjects will be blinded to treatment allocation. Ancef 1gm, or in the case of penicillin allergy, cipro 400 mg, will be given by intravenous.

A local anaesthetic will be instilled at the end of the cystoscopy (40 ml 1% lidocaine) and sedation will be provided as required. Fifteen minutes will lapse before beginning the procedure.

Using a 30 degree rigid scope and minimally invasive cystoscopic technique, 10 injections at 10 U/ml per injection (altogether 100 U of BTA) will be injected into the bladder wall, sparing the trigone.3,4 Subjects assigned to the placebo condition will receive injections of a saline at a similar frequency as the BTA injections.

Subjects will be observed for 60 minutes post procedure and then discharged home. This is the standard protocol for other BTA procedures performed on an outpatient basis in the RQHR. Catheter supplies will be provided upon discharge.

Follow-up Schedule:

1. Four to Six Weeks Post-Procedure: The primary and secondary measures will be assessed.
2. Three Months post-procedure: The same procedures will be repeated as at the four-to-six week assessment.
3. Six Months post-procedure: The four-to-six week assessment will be performed, and symptoms of retention or residual since the last visit will be discussed. A cystoscopy will be performed to study culture/urinalysis, measure desire and capacity, and show incontinence. Study allocation will be revealed at six months, and BTA injection will be offered to subjects that had received the placebo.
4. Nine Months: The four-to-six week procedures are repeated.
5. Twelve Months: The four-to-six week procedures are repeated.

Potential Significance:

Current anticholinergic therapy for non neurogenic UUI has limitations. In addition to significant systemic side effects, studies have shown that only 50% of patients improve with anticholinergic therapy, and that improvement does not always involve continence. Thus, detrusor injection of BTA may be a safe and efficacious therapy for patients who have failed standard therapy with anticholinergic medication and allow for an improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, greater than 17 years of age
* Written informed consent has been obtained
* Ability to follow study instructions and likely to complete all required visits
* Written authorization for Use and Release of Health and Research Study Information has been obtained
* Subject meets the following criteria: clinical diagnosis of urinary urge incontinence with resistance to or intolerance of anticholinergic medication
* Anticholinergic medications allowed
* Willingness and ability to use self-catheterization if necessary

Exclusion Criteria:

* Uncontrolled clinically significant medical condition other than the condition under evaluation
* Known allergy or sensitivity to any of the components in the study medication
* Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study
* Concurrent participation in another investigational drug or device study
* Treatment with botulinum toxin of any serotype for urological condition prior to enrolment in study (if applicable)
* Any medical condition that may put the subject at increased risk with exposure to botulinum toxin A including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Symptomatic urinary retention or post-void residual of >200ml
* Anticoagulation therapy within 3 days of injection procedure
* Familial bleeding disorder
* UUI secondary to neurologic disease
* Myasthenia gravis
* Previous bladder pathology (e.g. transitional cell carcinoma)

Ages: 17 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Jabs, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Kalsi V, Apostolidis A, Popat R, Gonzales G, Fowler CJ, Dasgupta P. Quality of life changes in patients with neurogenic versus idiopathic detrusor overactivity after intradetrusor injections of botulinum neurotoxin type A and correlations with lower urinary tract symptoms and urodynamic changes. Eur Urol. 2006 Mar;49(3):528-35. doi: 10.1016/j.eururo.2005.12.012. Epub 2006 Jan 6. PMID 16426735
- [Background] Sahai A, Khan MS, Dasgupta P. Efficacy of botulinum toxin-A for treating idiopathic detrusor overactivity: results from a single center, randomized, double-blind, placebo controlled trial. J Urol. 2007 Jun;177(6):2231-6. doi: 10.1016/j.juro.2007.01.130. PMID 17509328
- [Background] Sahai A, Kalsi V, Khan MS, Fowler CJ. Techniques for the intradetrusor administration of botulinum toxin. BJU Int. 2006 Apr;97(4):675-8. doi: 10.1111/j.1464-410X.2006.06063.x. No abstract available. PMID 16536751
- [Background] Rajkumar GN, Small DR, Mustafa AW, Conn G. A prospective study to evaluate the safety, tolerability, efficacy and durability of response of intravesical injection of botulinum toxin type A into detrusor muscle in patients with refractory idiopathic detrusor overactivity. BJU Int. 2005 Oct;96(6):848-52. doi: 10.1111/j.1464-410X.2005.05725.x. PMID 16153215
- [Background] Schurch B, de Seze M, Denys P, Chartier-Kastler E, Haab F, Everaert K, Plante P, Perrouin-Verbe B, Kumar C, Fraczek S, Brin MF; Botox Detrusor Hyperreflexia Study Team. Botulinum toxin type a is a safe and effective treatment for neurogenic urinary incontinence: results of a single treatment, randomized, placebo controlled 6-month study. J Urol. 2005 Jul;174(1):196-200. doi: 10.1097/01.ju.0000162035.73977.1c. PMID 15947626
- [Background] Vo AH, Satori R, Jabbari B, Green J, Killgore WD, Labutta R, Campbell WW. Botulinum toxin type-a in the prevention of migraine: a double-blind controlled trial. Aviat Space Environ Med. 2007 May;78(5 Suppl):B113-8. PMID 17547312
- [Background] Patki PS, Hamid R, Arumugam K, Shah PJ, Craggs M. Botulinum toxin-type A in the treatment of drug-resistant neurogenic detrusor overactivity secondary to traumatic spinal cord injury. BJU Int. 2006 Jul;98(1):77-82. doi: 10.1111/j.1464-410X.2006.06192.x. PMID 16831148
- [Background] Smith CP, Nishiguchi J, O'Leary M, Yoshimura N, Chancellor MB. Single-institution experience in 110 patients with botulinum toxin A injection into bladder or urethra. Urology. 2005 Jan;65(1):37-41. doi: 10.1016/j.urology.2004.08.016. PMID 15667859
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Nixon A, Colman S, Sabounjian L, Sandage B, Schwiderski UE, Staskin DR, Zinner N. A validated patient reported measure of urinary urgency severity in overactive bladder for use in clinical trials. J Urol. 2005 Aug;174(2):604-7. doi: 10.1097/01.ju.0000165461.38088.7b. PMID 16006914

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: normal saline injected into the detrusor in 5 sites on each side of the bladder (1 mL at each site) during cystoscopy
- Botulinum Toxin Type A: Botulinum toxin Type A 100U injected into the detrusor in 5 sites on each side of the bladder (1 mL at each site) during cystoscopy
Period: Overall Study
Arm/Group | Placebo | Botulinum Toxin Type A
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo injected into the detrusor at Day 1,
  Placebo: Placebo injected into the detrusor at Day 1, followed by injection of botulinum toxin Type A 100U after 24 weeks has elapsed from previous treatment, if requested/qualified.
- Botulinum Toxin Type A: Botulinum toxin Type A 100U injected into the detrusor at Day 1
  botulinum toxin Type A: Botulinum toxin Type A 100U injected into the detrusor at Day 1
- Total: Total of all reporting groups
Arm/Group | Placebo | Botulinum Toxin Type A | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.2) | 63 (9.4) | 63.38 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Capacity at Cystoscopy Between Baseline and 6 Month Follow-up
Description: Cystoscopy is a test performed with a cystoscope, a narrow tube with a tiny camera at its tip, inserted into the urethra and bladder to see the inside of the bladder and urethra.
  Maximum bladder capacity--the amount of liquid or gas the bladder can hold under anesthesia. Without anesthesia, capacity is limited by either pain or a severe urge to urinate.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
mL | -97.5 (176.92) | 64.1 (105.16)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; A sample of 16 subjects per group was required to detect a mean difference of 50 mL in maximum capacity at cystoscopy between botulinum toxin and placebo at 90% power with a two-sided type I error of 5%. Difference scores were computed for the primary outcome, which were then compared using the Wilcoxon- Mann-Whitney U test. This type of analysis was used to identify both between group differences and within group differences (over time) while using non-parametric statistics; Test type: Superiority or Other; p = .016, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

2. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 6 Week Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of episodes | .50 (1.75) | 3.00 (4.90)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.152, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

3. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 3 Month Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline to 3 month
Measure: Mean (Standard Deviation); unit: number of occurences
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of occurences | 1.28 (2.43) | 5.05 (5.06)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.095, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

4. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 6 Month Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline to 6 month
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of episodes | -.39 (3.58) | 4.09 (5.29)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.067, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

5. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 9 Month Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline to 9 months
Measure: Mean (Standard Deviation); unit: number of occurences
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of occurences | -3.38 (2.43) | NA (NA) — Data was not collected from this time period for the experimental group.

6. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 12 Month Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: number of occurences
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of occurences | -3.83 (2.06) | -2.17 (5.02)

7. Secondary Outcome: Change in Incontinence Episodes Between Baseline and 24 Months Follow-up
Description: Incontinence- involuntary leakage of urine
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: number of occurences
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of occurences | -3.75 (1.81) | -2.78 (7.55)

8. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 6 Week Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -0.50 (2.15) | 2.14 (2.55)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

9. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 3 Month Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 3 month
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | 0.89 (2.55) | 3.32 (3.09)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.095, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

10. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 6 Month Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -0.22 (2.39) | 2.73 (2.93)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.038, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

11. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 9 Month Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 9 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -1.13 (1.69) | NA (NA) — Data was not collected from this time period for the experimental group.

12. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 12 Month Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -1.61 (1.85) | -1.67 (2.36)

13. Secondary Outcome: Change in Number of Daytime Voids Between Baseline and 24 Month Follow-up
Description: Frequency of daily urination
Time Frame: Baseline to 24 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -0.33 (3.92) | -2.61 (2.85)

14. Secondary Outcome: Change in Number of Night Voids Between Baseline and 6 Week Follow-up
Description: Frequency of night voiding
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | 0.31 (1.31) | 0.77 (1.88)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.904, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

15. Secondary Outcome: Change in Number of Night Voids Between Baseline and 3 Month Follow-up
Description: Frequency of night voiding
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: Number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
Number of voids | 0.06 (1.29) | 1.36 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.080, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

16. Secondary Outcome: Change in Number of Night Voids Between Baseline and 6 Month Follow-up
Description: Frequency of night voiding
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | 0.33 (0.79) | 1.32 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.230, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

17. Secondary Outcome: Change in Number of Night Voids Between Baseline and 9 Month Follow-up
Description: Frequency of night voiding
Time Frame: Baseline and 9 months
Measure: Mean (Standard Deviation); unit: Number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
Number of voids | -1.13 (1.03) | NA (NA) — Data was not collected from this time period for the experimental group.

18. Secondary Outcome: Change in Number of Night Voids Between Baseline and 12 Month Follow-up
Description: Frequency of night voiding
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -0.94 (1.16) | -1.28 (1.33)

19. Secondary Outcome: Change in Number of Night Voids Between Baseline and 24 Months Follow-up
Description: Frequency of night voiding
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: number of voids
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of voids | -0.72 (1.25) | -1.00 (1.35)

20. Secondary Outcome: Subjective Benefit Assessment at 6 Weeks
Description: Self assessed description of how well they believed the Botulinum Toxin type A was working. The patients' subjective assessment of the treatment's efficacy was obtained verbally using a four-point rating scale. Rating options were:
  1. dry (complete response),
  2. improvement (> 50% reduction in incontinence),
  3. partial response (≤ 50% reduction in incontinence),
  4. no response to treatment.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a 4-point rating scale
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
score on a 4-point rating scale | 3.4 (0.9) | 2.4 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.1 to -0.2]

21. Secondary Outcome: Subjective Benefit Assessment at 3 Months
Description: as for outcome 20
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a 4-point rating scale
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
score on a 4-point rating scale | 3.2 (0.9) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.1 to -0.5]

22. Secondary Outcome: Subjective Benefit Assessment at 6 Months
Description: Self assessed description of how well they believed the Botulinum Toxin type A was working.The patients' subjective assessment of the treatment's efficacy was obtained verbally using a four-point rating scale. Rating options were:
  1. dry (complete response),
  2. improvement (> 50% reduction in incontinence),
  3. partial response (≤ 50% reduction in incontinence),
  4. no response to treatment.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: score on a 4-point rating scale
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
score on a 4-point rating scale | 2.8 (0.9) | 1.6 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-2.0 to -0.4]

23. Secondary Outcome: Change in Incontinence Impact Questionnaire From Baseline to 6 Weeks Follow-up
Description: Disease specific validated quality of life measure. Health-related quality of life measures for women with urinary incontinence.
  Incontinences Impact Questionnaire - 7 (IIQ-7) The IIQ-7 is 7-point scale used to rate a patients' life and the affect of accidental urine loss on activities, relationships, and feelings. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
scores on a scale | .00 (14.02) | 27.27 (41.51)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.173, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

24. Secondary Outcome: Change in Incontinence Impact Questionnaire From Baseline to 3 Months Follow-up
Description: as for outcome 23
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 4.29 (15.30) | 35.35 (41.19)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.051, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

25. Secondary Outcome: Change in Incontinence Impact Questionnaire From Baseline to 6 Months Follow-up
Description: as for outcome 23
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 3.81 (33.95) | 34.63 (36.76)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.051, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

26. Secondary Outcome: Change in Urogenital Distress Inventory From Baseline to 6 Week Follow-up
Description: Disease specific quality of life measure. Health-related quality of life measures for women with urinary incontinence.
  Urogenital Distress Inventory - 6 (UDI-6) The UDI-6 is a 6-point scale that asks patients to respond to questions rating whether they experience and how much they are bothered by UUI. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. Higher scores reflect greater distress associated with symptoms. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 6.11 (15.37) | 17.68 (30.20)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.557, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

27. Secondary Outcome: Change in Urogenital Distress Inventory From Baseline to 3 Months Follow-up
Description: Disease specific quality of life measure. Health-related quality of life measures for women with urinary incontinence.
  The UDI-6 is a 6-point scale that asks patients to respond to questions rating whether they experience and how much they are bothered by UUI. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. Higher scores reflect greater distress associated with symptoms. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 15.33 (14.44) | 32.32 (19.69)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.029, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

28. Secondary Outcome: Change in Urogenital Distress Inventory From Baseline to 6 Months Follow-up
Description: as for outcome 27
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 11.11 (23.57) | 28.48 (17.41)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.132, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

29. Secondary Outcome: Change in Patient Perception of Bladder Condition From Baseline to 6 Weeks
Description: Disease specific validated quality of life measures. A single-item global measure for patients with overactive bladder.
  Patient Perception of Bladder Condition (PPBC) The PPBC is a single-item, 6-point scale that asks patients to rate their subjective impression of their current bladder problems. It has been shown to have concurrent and discriminant validity as well as responsiveness to treatment. Patients are asked to rate their perceived bladder condition on a 6-point scale ranging from 1 "no problems at all", 2 "some very minor problems". 3 "some minor problems", 4"(some) moderate problems", 5 "severe problems", and 6 "many severe problems". A higher score indicates a more negative impression of current bladder problems.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | .20 (.79) | 1.45 (1.75)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.085, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

30. Secondary Outcome: Change in Patient Perception of Bladder Condition From Baseline to 3 Months
Description: as for outcome 29
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | .50 (1.27) | 1.82 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.099, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

31. Secondary Outcome: Change in Patient Perception of Bladder Condition From Baseline to 6 Months
Description: as for outcome 29
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | .50 (1.43) | 1.55 (1.75)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.132, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

32. Secondary Outcome: Change in Indevus Urgency Severity Scale From Baseline to 6 Weeks
Description: A disease specific quality of life measure. A self reported measure that assesses urinary urgency severity associated with overactive bladder.
  Indevus Urgency Severity Scale (IIUS) The IIUS is a single item scale designed to describe urinary urges. The scale is rated through the patient's urge: none (0 points), mild (1), moderate (2) and severe (3). A higher score represents more urinary urges.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 1.00 (0.88) | 1.09 (1.30)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.072, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

33. Secondary Outcome: Change in Indevus Urgency Severity Scale From Baseline to 3 Months
Description: as for outcome 32
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 0.67 (1.0) | 1.36 (1.12)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.230, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

34. Secondary Outcome: Change in Indevus Urgency Severity Scale From Baseline to 6 Months
Description: as for outcome 32
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: summary score
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
summary score | 0.60 (0.97) | 1.09 (.94)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.314, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

35. Secondary Outcome: 24 Hour Pad Weight (gm) at 3 Months
Description: weight of pad (in gm) worn for 24 hours to detect urine loss
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
gm | 413.30 (558.82) | 141.18 (301.93)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.013, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

36. Secondary Outcome: 24 Hour Pad Weight (gm) at 9 Months
Description: weight of pad (in gm) worn for 24 hours to detect urine loss
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: gm
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
gm | 64.11 (145.36) | 110.63 (277.01)
Statistical Analysis 1: Comparison: Placebo vs Botulinum Toxin Type A; Test type: Superiority or Other; p = 0.888, Wilcoxon (Mann-Whitney); A Bonferroni correction (0.05/n) was used for multiple comparisons

37. Secondary Outcome: Frequency of Urinary Tract Infections From Baseline to 6 Months
Description: Frequency of urinary tract infections from baseline to 6 month-follow-up
Time Frame: Baseline to 6 months
Measure: Number; unit: number of occurences
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
number of occurences | 4 | 6

38. Secondary Outcome: Frequency of Participants Needing Self-catheterization From Baseline to 6 Month Follow-up
Description: Frequency of participants needing self-catheterization from baseline to 6 month follow-up.
Time Frame: Baseline to 6 months
Measure: Number; unit: Participants
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
Participants | 0 | 1

39. Secondary Outcome: Frequency of Participants With Urinary Tract Infections From Baseline to 6 Months
Description: Frequency of particiapnts with urinary tract infections from baseline to 6 month-follow-up
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Botulinum Toxin Type A
Number analyzed (Participants) | 10 | 11
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline up to 12 months after intervention (at 4-6 weeks, 3 months, 6 months, 9 months and 12 months).
Arm/Group | Placebo | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/11
Other Adverse Events (participants affected / at risk) | 3/10 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Botulinum Toxin Type A (N=11)
Perioperative Cardiac Event (Takotsubo syndrome) (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Botulinum Toxin Type A (N=11)
Hematuria (Infections and infestations) | 1 | 1
Pain/Discomfort (General disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Poor recruitment. Recruitment slowed significantly when newer anticholinergic medications became available. Those who were previously eligible for the study had darifenacin and solifenacin to try before considering botulinum toxin treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes